CLINICAL TRIAL: NCT04377360
Title: A Pilot Feasibility Trial of Diffusing Alpha-emitter Radiation Therapy (DaRT) for Malignant Skin and Superficial Soft Tissue Tumors
Brief Title: Feasibility Trial of Diffusing Alpha-emitter Radiation Therapy (DaRT) for Malignant Skin & Superficial Soft Tissue Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-SCC-MSK-00
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-07

CONDITIONS: Malignant Skin Tumor; Soft Tissue Tumor, Malignant
Keywords: Skin Tumor; Superficial Soft Tissue Tumor
MeSH Terms: conditions — Skin Neoplasms; Sarcoma

STUDY DESIGN:
Intervention Model Description: This is a multi-center feasibility trial with DaRT for the treatment of malignant skin and superficial soft tissue tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Diffusing Alpha-emitter Radiation Therapy (DaRT) (Experimental): DaRT source will be inserted using preplanned radiotherapy parameters and reassessed by volumetric imaging 2-3 weeks after placement and then removed. Tumor response to DaRT will be assessed periodically 3 months after removal.
  Interventions: Radiation: Diffusing Alpha-emitter Radiation Therapy

INTERVENTIONS:
Radiation: Diffusing Alpha-emitter Radiation Therapy — Diffusing Alpha-emitter Radiation Therapy (DaRT) is a method of delivering interstitial brachytherapy, based on the interstitial intratumoral placement of an encapsulated Radium-224 source (3.7 days half-life). These sources release short-lived alpha-emitting atoms into the tumor microenvironment by recoil. As the radioisotope has a short half-life, the majority of radiation absorption happens in the tumor.
  Other Names: DaRT

SUMMARY:
This is a single-institution pilot feasibility trial in which 10 subjects will be enrolled. The primary objectives are is to explore the feasibility of delivering radiotherapy for malignant skin and superficial soft tissue tumors using DaRT (Alpha Tau Medical, Tel Aviv, Israel), a form of interstitial brachytherapy which uses a novel radioisotope delivery system, as well as to determine the frequency and severity of acute adverse events. Secondary objectives will include assessments of radiotherapy-related adverse events, tumor response, radiation safety, stability of device placement, and associations with quality of life.

DETAILED DESCRIPTION:
Diffusing Alpha-emitter Radiation Therapy is a form of interstitial brachytherapy which may be effective in treating malignant skin and superficial soft tissue tumors for several reasons. First, alpha-emitting radionuclides have a high linear energy transfer (LET), which produces a dense track of ionization events within cells and DNA, which produce complex DNA damage and more effective cell kill than more sparsely ionizing forms of radiation, such as gamma-rays or x-rays. Second, alpha-emitting radionuclides exhibit a higher relative biologic effect (RBE) compared to gamma-rays or x-rays, due to the relative insensitivity to cancer cellular radiosensitivity associated with cell cycling. Finally, alpha-emitting radionuclides are relatively insensitive to hypoxia, which is common as malignant skin and superficial soft tissue tumors become larger (Hall 2000).

Alpha particles have been considered unsuitable for treatment of solid tumors, since no practical method to effectively irradiate a macroscopic tumor with these short-range particles (penetration range in human tissue of ≤0.1 mm) has been found.

The "Diffusing Alpha-emitter Radiation Therapy (DaRT)", based on the interstitial intratumoral placement of an encapsulated Radium-224 source (3.7 days half-life), is described in this study. These sources release short-lived alpha-emitting atoms into the tumor microenvironment by recoil. These atoms are dispersed in the immediate surrounding tumor microenvironment both by convection through tumor interstitial fluid and by thermal diffusion. The decay of Radium-224 in the capsule results in the release of the short-lived (half-life of about 1 minute) radioisotope Radon-220. Radon-220 migrates in the tumor microenvironment until it decays. This is followed by the decay of its daughter radioisotope, Polonium-216. Lead-212, the result of this last decay, gives rise to Bismuth-212, which emits yet another alpha particle. The result of these decay events is the release of alpha particles (Kelson 1994 and Kelson 1995). DaRT will be used in this study for the treatment of malignant skin and superficial soft tissue tumors.

This study has been designed to determine the feasibility of performing the procedure required to deliver radiotherapy to the tumor. At the same time, the safety of the treatment, tumor response, radiation safety, device placement stability, and patient reported quality of life, and molecular and histologic effects on the tumor will be assessed.

The DaRT sources will be inserted using preplanned radiotherapy parameters, with a specified number and size of DaRT sources. Approximately 2-3 weeks after placement of the DaRT sources, the placement of the sources will be reassessed by volumetric imaging, and then they will be removed. Tumor response to DaRT will be assessed periodically 3 months after removal of the device.

This is a single-institution pilot feasibility trial in which 10 subjects will be enrolled.

The primary objectives are is to explore the feasibility of delivering radiotherapy for malignant skin and superficial soft tissue tumors using DaRT (Alpha Tau Medical, Tel Aviv, Israel), a form of interstitial brachytherapy which uses a novel radioisotope delivery system, as well as to determine the frequency and severity of acute adverse events. Secondary objectives will include assessments of radiotherapy-related adverse events, tumor response, radiation safety, stability of device placement, and associations with quality of life.

ELIGIBILITY:
* Malignant tumor of the skin or superficial soft tissue*, ≥10 mm and ≤50 mm in longest dimension, with minimum tumor thickness of 4 mm
* *Including, but after review by the Principal Investigator not limited to:

  * Primary malignant tumors of the skin such as keratinocytic carcinomas (basal cell carcinoma, squamous cell carcinoma), melanocytic tumors (melanoma), soft tissue tumors (cutaneous angiosarcoma or leiomyosarcoma), and neural tumors (Merkel cell carcinoma)
  * Primary malignant tumors of the superficial soft tissues such as adipocytic tumors (liposarcoma), smooth-muscle tumors (leiomyosarcoma), skeletal muscle tumors (rhabdomyosarcoma), vascular tumors (Kaposi sarcoma, angiosarcoma of soft tissue)
  * Secondary malignant tumors of the skin and superficial soft tissues such as metastases from breast cancer, lung cancer, melanoma, kidney cancer and others.
* Limited treatment options for the tumor, including:

  * Recurrent tumors that must have failed at least one standard therapy, which includes previous radiotherapy or surgery, OR
  * Tumors in patients with metastases who will not be rendered disease-free by tumor resection, OR
  * Tumors deemed inappropriate for resection by a surgeon for one of the following reasons:

    * Complete tumor resection unlikely because of tumor location or size;
    * Complete tumor resection deemed excessively morbid or deforming (e.g., requiring amputation of digit, lip, eyelid, ear);
    * Patient with medical comorbidity contraindicating surgery; or
    * Patent refusal due to anticipated morbidity
* Age >18 years
* Eastern cooperative oncology group performance status ≤3
* Life expectancy ≥12 weeks
* Platelet count ≥50,000/mm3
* International normalized ratio of prothrombin time ≤1.8
* Creatinine ≤1.9 mg/dL

Subject Exclusion Criteria

* Contraindication to radiotherapy for skin and superficial soft tissue tumor
* Radiotherapy to the malignant skin or soft tissue tumor planned for radiotherapy within last 6 months
* Prior radiotherapy to the malignant skin or soft tissue tumor planned for radiotherapy with doses > 60 Gy (equivalent dose in 2 Gy fractions using α/β of 8.5)
* Anticoagulation or antiplatelet medical therapy
* High probability of non-compliance with scheduled assessments as demonstrated by prior inability to complete scheduled routine clinical assessments
* Pregnancy
* Women of childbearing potential unwilling or unable to use an acceptable contraceptive method to prevent pregnancy for 1 year after brachytherapy
* Men unwilling or unable to use an acceptable contraceptive method to prevent pregnancy for 1 year after brachytherapy
* Inability to read or understand English (as QoL questionnaires are only validated in English)
* Concurrent receipt of cancer therapy which has proven effective for the malignant skin or soft tissue tumor planned for radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of DaRT Delivery | 1 Day
  To explore feasibility of delivering radiotherapy for malignant skin and superficial soft tissue tumors using Diffusing Alpha-emitter Radiation Therapy (DaRT). Feasibility will be determined by successful delivery of radiation by DaRT to the malignant tumor. If an attempt to place the DaRT is unsuccessful, this patient will be considered a feasibility failure. A feasibility failure may be due to inability to execute the workflow of pre-brachytherapy imaging, treatment planning, device procurement, or technical inability to place the DaRT sources into the skin and superficial soft tissue tumor. The rate of feasibility failures will be reported.
Frequency and Severity of Adverse Events | Up to 24 Weeks after DaRT Removal
  To determine the frequency and severity of acute adverse events related to DaRT for skin and superficial soft tissue tumors. Adverse events will be assessed and graded according to Common Terminology and Criteria for adverse events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Rate of Tumor Response using Response Evaluation Criteria in Solid Tumors (RECIST) | 3 Months
  To assess the rate of malignant skin and superficial soft tissue tumor response after DaRT. Tumor response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 using calibrated digital photography and CT imaging 3 months after DaRT.
Radiation Exposure Safety using a Calibrated Survey Probe | 1 Day
  To assess radiation safety through determination of patient and personnel radiation exposure during DaRT. Radiation exposure will be measured using a calibrated survey probe.
Stability Assessment of the DaRT Sources after Placement | 2 Weeks
  To assess stability of the DaRT sources after placement. Stability will be assessed by localization of the DaRT sources in the tumor after placement, measured by geometric comparisons of the DaRT sources relative to the centroid of the tumor, using brachytherapy planning software. Distance of the DaRT sources relative to the centroid immediately at the time of initial placement and immediately before removal will be analyzed and reported numerically.
Quality of Life Assessment using the Skindex-16 | 2 Weeks after DaRT Placement and 6, 12, 24 Weeks after DaRT Removal
  To assess skin-related and cancer-related quality of life (QoL) after DaRT. QoL will be assessed using the Skindex-16 following placement of the DaRT. The Skindex-16 scores range from 0 to 100 (with higher scores representing lower satisfaction).
Quality of Life Assessment using the Skin Cancer Index (SCI) | 2 Weeks after DaRT Placement and 6, 12, 24 Weeks after DaRT Removal
  To assess skin-related and cancer-related quality of life (QoL) after DaRT. QoL will be assessed using the Skin Cancer Index (SCI) following placement of the DaRT. The SCI scores range from 5-22 (with higher scores indicating higher QOL).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - UnityPoint Health - John Stoddard Cancer Center, Des Moines, Iowa
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - University Cancer & Diagnostic Center, Houston, Texas
  - Dermatology of Seattle and Bellevue, Seattle, Washington

REFERENCES:
- [Derived] D'Andrea MA, VanderWalde NA, Ballo MT, Patra P, Cohen GN, Damato AL, Barker CA. Feasibility and Safety of Diffusing Alpha-Emitter Radiation Therapy for Recurrent or Unresectable Skin Cancers. JAMA Netw Open. 2023 May 1;6(5):e2312824. doi: 10.1001/jamanetworkopen.2023.12824. PMID 37166798